CLINICAL TRIAL: NCT00920218
Title: Safety and Immunogenicity of GlaxoSmithKline Biologicals' Herpes Zoster Vaccine 1437173A
Brief Title: Safety & Immunogenicity of GlaxoSmithKline Biologicals' Herpes Zoster Vaccine 1437173A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 110258
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-08

CONDITIONS: Herpes Zoster
Keywords: Vaccine; Safety; Herpes Zoster; Immunogenicity; Stem cell transplantation
MeSH Terms: conditions — Herpes Zoster | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- GSK 1437173A F1 Group (Experimental): Male or female subjects, 18 years of age or older at the time of the first vaccination, received 3 doses of GSK 1437173A formulation 1 (F1) vaccine, administered intramuscularly in the upper deltoid region of non-dominant arm according to a 0,1,3-months schedule.
  Interventions: Biological: Herpes Zoster Vaccine 1437173A
- GSK 1437173A F2 Group (Experimental): Male or female subjects, 18 years of age or older at the time of the first vaccination, received 3 doses of GSK 1437173A formulation 2 (F2) vaccine, administered intramuscularly in the upper deltoid region of non-dominant arm according to a 0,1,3-months schedule.
  Interventions: Biological: Herpes Zoster Vaccine 1437173A
- Placebo-GSK 1437173A F1 Group (Experimental): Male or female subjects, 18 years of age or older at the time of the first vaccination, received 1 dose of the placebo followed by 2 doses of GSK 1437173A F1 vaccine. For some safety analyses, this Group was split into Placebo 1D Group (results following placebo administration) and GSK 1437173A 2D Group (results following HZV administration). All vaccines were administered intramuscularly in the upper deltoid region of non-dominant arm according to a 0,1,3-months schedule.
  Interventions: Biological: Herpes Zoster Vaccine 1437173A; Biological: Placebo vaccine (saline)
- Placebo Group (Placebo Comparator): Male or female subjects, 18 years of age or older at the time of the first vaccination, received 3 doses of placebo, administered intramuscularly in the upper deltoid region of non-dominant arm according to a 0,1,3-months schedule.
  Interventions: Biological: Placebo vaccine (saline)

INTERVENTIONS:
Biological: Herpes Zoster Vaccine 1437173A — Different formulations of investigational vaccine (GSK 1437173A) administered in 2 or 3 doses intramuscularly.
  Arms: GSK 1437173A F1 Group; GSK 1437173A F2 Group; Placebo-GSK 1437173A F1 Group
Biological: Placebo vaccine (saline) — 1 or 3 doses of Placebo (saline) injected intramuscularly.
  Arms: Placebo Group; Placebo-GSK 1437173A F1 Group

SUMMARY:
The purpose of this observer-blind study is to evaluate the safety and immunogenicity of GlaxoSmithKline Biologicals' investigational Herpes Zoster vaccine GSK1437173A when administered as 2 doses or 3 doses to hematopoietic stem cell transplant (HCT) recipients.

DETAILED DESCRIPTION:
The Protocol Posting has been updated following Protocol amendment 2, Sep 2009. The sections impacted are: eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol;
* Male and female subjects at least 18 years old at the time of vaccination;
* Serological evidence of prior VZV infection for all subjects born in 1980 or later and for subjects born outside the US before 1980 in a tropical or sub-tropical region. No testing for serological evidence of prior VZV infection is required for US subjects born before 1980;
* Has undergone autologous HCT within the past 50-70 days for treatment of Hodgkin lymphoma, non-Hodgkin lymphoma (T or B cell), myeloma or acute myeloid leukemia, and there are no plans for additional HCTs
* Written informed consent obtained from the subject;
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period;
* Administration or planned administration of a vaccine that is not part of the study protocol since transplantation. However licensed non-replicating vaccines (i.e. inactivated and subunit vaccines, including inactivated and subunit influenza vaccines, with or without adjuvant) may be administered up to 8 days prior to dose 1;
* Administration of immunoglobulins since transplantation;
* Previous vaccination against varicella or HZ;
* History of HZ within the previous 12 months;
* Known exposure to VZV since transplantation;
* Evidence of active infection at the time of enrollment including a temperature of ≥ 37.5° C or any serious HCT-related complication;
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine;
* Hypersensitivity or intolerance to acyclovir or valacyclovir;
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-07-14 (Actual); Primary Completion 2011-04-26 (Actual); Study Completion 2012-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneota, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Stadtmauer EA, Sullivan KM, Marty FM, Dadwal SS, Papanicolaou GA, Shea TC, Mossad SB, Andreadis C, Young JA, Buadi FK, El Idrissi M, Heineman TC, Berkowitz EM. A phase 1/2 study of an adjuvanted varicella-zoster virus subunit vaccine in autologous hematopoietic cell transplant recipients. Blood. 2014 Nov 6;124(19):2921-9. doi: 10.1182/blood-2014-04-573048. Epub 2014 Sep 18. PMID 25237196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Serological evidence of prior Varicella-Zoster Virus infection for those born in 1980 or later and for those born outside the US before 1980 in a tropical or sub-tropical region was required. All subjects were to have undergone autologous hematopoietic stem cell transplantation (HCT) within the past 50-70 days; and had no additional HCTs planned.
Pre-assignment Details: Out of the 121 subjects enrolled into this study, 1 subject was eliminated due to not receiving study vaccination and hence only 120 subjects started.
Period: Overall Study
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Started | 30 | 29 | 31 | 30
Completed | 28 | 24 | 23 | 23
Not Completed | 2 | 5 | 8 | 7
Not completed — Serious Adverse Event | 2 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 3
Not completed — Transplant failed/malignancy recurrence | 0 | 1 | 2 | 3
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group | Total
Number analyzed (Participants) | 30 | 29 | 31 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (12.2) | 56.0 (11.4) | 57.8 (6.8) | 57.3 (8.6) | 56.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 10 | 11 | 42
  Male | 18 | 20 | 21 | 19 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African Heritage/African American | 2 | 2 | 1 | 1 | 6
  Race/Ethnicity: American Indian or Alaskan Native | 0 | 1 | 0 | 0 | 1
  Race/Ethnicity: Asian-Central/South Asian Heritage | 0 | 0 | 0 | 1 | 1
  Race/Ethnicity: Asian-East Asian Heritage | 0 | 0 | 0 | 2 | 2
  Race/Ethnicity: Asian-Japanese Heritage | 1 | 0 | 0 | 0 | 1
  Race/Ethnicity: Other | 2 | 2 | 0 | 4 | 8
  Race/Ethnicity: White-Arabic/North African Heritage | 1 | 0 | 0 | 0 | 1
  Race/Ethnicity: White-Caucasian/European Heritage | 24 | 24 | 30 | 22 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-days (Days 0-6) post-vaccination period following each dose and across doses
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Groups:
- GSK 1437173A 2D Group: Subgroup of Placebo-GSK 1437173A F1 Group, results following GSK 1437173A vaccine administration.
- Placebo 1D Group: Subgroup of Placebo-GSK 1437173A F1 Group, results following placebo administration.
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | GSK 1437173A 2D Group | Placebo 1D Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 28 | 30 | 30
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Pain, Dose 1 | 25 | 19 | 22 | 4 | 3
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Pain, Dose 1 | 0 | 3 | 1 | 0 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Redness, Dose 1 | 2 | 6 | 2 | 1 | 0
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Swelling, Dose 1 | 1 | 3 | 4 | 0 | 0
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Pain, Dose 2 | 24 | 19 | 22 |  | 3
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Pain, Dose 2 | 2 | 3 | 1 |  | 0
  Any Redness, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Redness, Dose 2 | 2 | 2 | 7 |  | 1
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 |  | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Swelling, Dose 2 | 1 | 1 | 3 |  | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 |  | 0
  Any Pain, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 23
  Any Pain, Dose 3 | 24 | 15 |  |  | 4
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 23
  Grade 3 Pain, Dose 3 | 1 | 0 |  |  | 0
  Any Redness, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 23
  Any Redness, Dose 3 | 6 | 4 |  |  | 0
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 23
  Grade 3 Redness, Dose 3 | 0 | 0 |  |  | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 23
  Any Swelling, Dose 3 | 4 | 1 |  |  | 0
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 23
  Grade 3 Swelling, Dose 3 | 0 | 0 |  |  | 0
  Any Pain, Across Doses | 27 | 22 | 24 | 4 | 7
  Grade 3 Pain, Across Doses | 3 | 5 | 1 | 0 | 0
  Any Redness, Across Doses | 6 | 7 | 7 | 1 | 1
  Grade 3 Redness, Across Doses | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across Doses | 6 | 4 | 4 | 0 | 0
  Grade 3 Swelling, Across Doses | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms [including nausea, vomiting, diarrhoea and abdominal pain], temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache and myalgia. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = temperature higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-days (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | GSK 1437173A 2D Group | Placebo 1D Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 28 | 30 | 30
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Fatigue, Dose 1 | 13 | 11 | 12 | 15 | 7
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Fatigue, Dose 1 | 1 | 1 | 0 | 1 | 0
  Related Fatigue, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Related Fatigue, Dose 1 | 5 | 7 | 8 | 6 | 1
  Any Gastr. sympt., Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Gastr. sympt., Dose 1 | 6 | 4 | 1 | 9 | 2
  Grade 3 Gastr. sympt., Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Gastr. sympt., Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Gastr. sympt., Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Related Gastr. sympt., Dose 1 | 3 | 2 | 1 | 3 | 1
  Any Headache, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Headache, Dose 1 | 4 | 1 | 4 | 7 | 2
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Headache, Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Headache, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Related Headache, Dose 1 | 3 | 1 | 4 | 2 | 1
  Any Myalgia, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Myalgia, Dose 1 | 14 | 12 | 13 | 9 | 3
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Myalgia, Dose 1 | 1 | 0 | 1 | 0 | 0
  Related Myalgia, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Related Myalgia, Dose 1 | 12 | 9 | 10 | 6 | 2
  Any Temperature, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Any Temperature, Dose 1 | 3 | 3 | 5 | 7 | 1
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 2 | 0
  Related Temperature, Dose 1: number analyzed (Participants) | 30 | 29 | 27 | 30 | 30
  Related Temperature, Dose 1 | 3 | 2 | 4 | 5 | 1
  Any Fatigue, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Fatigue, Dose 2 | 10 | 8 | 16 |  | 8
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Fatigue, Dose 2 | 3 | 1 | 1 |  | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Related Fatigue, Dose 2 | 7 | 3 | 10 |  | 3
  Any Gastr. sympt., Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Gastr. sympt., Dose 2 | 2 | 2 | 6 |  | 2
  Grade 3 Gastr. sympt., Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Gastr. sympt., Dose 2 | 0 | 0 | 1 |  | 0
  Related Gastr. sympt., Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Related Gastr. sympt., Dose 2 | 1 | 2 | 2 |  | 0
  Any Headache, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Headache, Dose 2 | 7 | 1 | 6 |  | 2
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Headache, Dose 2 | 2 | 0 | 0 |  | 0
  Related Headache, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Related Headache, Dose 2 | 4 | 0 | 4 |  | 1
  Any Myalgia, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Myalgia, Dose 2 | 13 | 13 | 19 |  | 5
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Myalgia, Dose 2 | 4 | 2 | 1 |  | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Related Myalgia, Dose 2 | 12 | 11 | 12 |  | 3
  Any Temperature, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Any Temperature, Dose 2 | 10 | 4 | 4 |  | 1
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0 |  | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 29 | 27 | 26 | 0 | 29
  Related Temperature, Dose 2 | 8 | 3 | 4 |  | 0
  Any Fatigue, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Any Fatigue, Dose 3 | 15 | 10 |  |  | 8
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Grade 3 Fatigue, Dose 3 | 3 | 0 |  |  | 1
  Related Fatigue, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Related Fatigue, Dose 3 | 9 | 8 |  |  | 3
  Any Gastr. sympt., Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Any Gastr. sympt., Dose 3 | 9 | 5 |  |  | 2
  Grade 3 Gastr. sympt., Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Grade 3 Gastr. sympt., Dose 3 | 0 | 0 |  |  | 0
  Related Gastr. sympt., Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Related Gastr. sympt., Dose 3 | 4 | 3 |  |  | 1
  Any Headache, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Any Headache, Dose 3 | 12 | 1 |  |  | 4
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Grade 3 Headache, Dose 3 | 2 | 0 |  |  | 0
  Related Headache, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Related Headache, Dose 3 | 9 | 1 |  |  | 3
  Any Myalgia, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Any Myalgia, Dose 3 | 18 | 7 |  |  | 5
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Grade 3 Myalgia, Dose 3 | 4 | 0 |  |  | 1
  Related Myalgia, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Related Myalgia, Dose 3 | 14 | 7 |  |  | 4
  Any Temperature, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Any Temperature, Dose 3 | 6 | 3 |  |  | 2
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Grade 3 Temperature, Dose 3 | 1 | 0 |  |  | 0
  Related Temperature, Dose 3: number analyzed (Participants) | 28 | 24 | 0 | 0 | 22
  Related Temperature, Dose 3 | 6 | 3 |  |  | 1
  Any Fatigue, Across Doses | 18 | 18 | 20 | 15 | 10
  Grade 3 Fatigue, Across Doses | 4 | 2 | 1 | 1 | 1
  Related Fatigue, Across Doses | 11 | 11 | 14 | 6 | 5
  Any Gastr. sympt., Across Doses | 10 | 7 | 6 | 9 | 4
  Grade 3 Gastr. sympt., Across Doses | 0 | 0 | 1 | 0 | 0
  Related Gastr. sympt., Across Doses | 7 | 5 | 2 | 3 | 2
  Any Headache, Across Doses | 13 | 3 | 9 | 7 | 6
  Grade 3 Headache, Across Doses | 3 | 0 | 0 | 0 | 0
  Related Headache, Across Doses | 9 | 2 | 7 | 2 | 5
  Any Myalgia, Across Doses | 21 | 18 | 22 | 9 | 8
  Grade 3 Myalgia, Across Doses | 8 | 2 | 1 | 0 | 1
  Related Myalgia, Across Doses | 19 | 15 | 16 | 6 | 5
  Any Temperature, Across Doses | 12 | 8 | 8 | 7 | 4
  Grade 3 Temperature, Across Doses | 1 | 0 | 0 | 2 | 0
  Related Temperature, Across Doses | 10 | 7 | 7 | 5 | 2

3. Primary Outcome: Number of Subjects With Any and Grade 3 Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | GSK 1437173A 2D Group | Placebo 1D Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 29 | 31 | 30
Participants
  Any AEs | 25 | 23 | 22 | 16 | 21
  Grade 3 AEs | 5 | 6 | 2 | 1 | 4

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Any time during the study up to Day 29 after the last vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | GSK 1437173A 2D Group | Placebo 1D Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 29 | 31 | 30
Participants | 3 | 5 | 2 | 1 | 2

5. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 4
Time Frame: During the entire study period (from Day 0 up to Month 15)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 31 | 30
Participants | 6 | 9 | 10 | 8

6. Primary Outcome: Number of Subjects With Any New Onset of Autoimmune Diseases (NOADs) and Other Immune Mediated Inflammatory Disorders
Description: Any new onset of autoimmune diseases and immune mediated inflammatory disorders were to be reported throughout the entire study period, whether or not they were considered to be possibly related to the treatment administration. These included neurological/demyelinating events, rheumatic and connective diseases, autoimmune endocrine diseases, inflammatory bowel diseases, autoimmune blood disorders, inflammatory skin disorders, other autoimmune/inflammatory events, autoimmune bullous skin diseases, vasculitis and liver autoimmune diseases.
Time Frame: Within the 30-day (Days 0-29) post last vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 31 | 30
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Any New Onset of Autoimmune Diseases (NOADs) and Other Immune Mediated Inflammatory Disorders
Description: as for outcome 6
Time Frame: During the entire study period (from Day 0 to Month 15)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 31 | 30
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Hematological and Biochemical Parameters With Respect to Normal Laboratory Ranges
Description: Hematological and biochemical parameters assessed were Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Basophils (BAS), Calcium (CAL), Creatinine (CREA), Eosinophils (EOS), Fibrinogen (FIBR), Hemoglobin (HGB), Hematocrit (HCT), Lactate Dehydrogenase (LDH), Lymphocytes (LYM), Monocytes (MON), Neutrophils (NEU), Platelets (PLAT), Prothrombin Time (PT), Partial Thromboplastin Time (PTT), Red Blood Cells (RBC), Total Protein (TP) and White Blood Cells (WBC).
Time Frame: At Month 0
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 31 | 30
Participants
  ALT: Unknown | 0 | 0 | 0 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 28 | 29 | 31 | 29
  ALT: Above | 2 | 0 | 0 | 1
  AST: Unknown | 0 | 0 | 1 | 1
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 29 | 29 | 29 | 28
  AST: Above | 1 | 0 | 1 | 1
  BAS: Unknown | 0 | 0 | 0 | 1
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 30 | 29 | 31 | 29
  BAS: Above | 0 | 0 | 0 | 0
  CAL: Unknown | 0 | 0 | 1 | 1
  CAL: Below | 0 | 2 | 1 | 3
  CAL: Normal | 30 | 27 | 29 | 26
  CAL: Above | 0 | 0 | 0 | 0
  CREA: Unknown | 0 | 0 | 0 | 0
  CREA: Below | 1 | 0 | 1 | 1
  CREA: Normal | 28 | 25 | 27 | 27
  CREA: Above | 1 | 4 | 3 | 2
  EOS: Unknown | 0 | 0 | 0 | 1
  EOS: Below | 5 | 1 | 6 | 6
  EOS: Normal | 24 | 28 | 23 | 21
  EOS: Above | 1 | 0 | 2 | 2
  FIBR: Unknown | 2 | 0 | 1 | 4
  FIBR: Below | 3 | 0 | 5 | 0
  FIBR: Normal | 25 | 22 | 21 | 24
  FIBR: Above | 0 | 7 | 4 | 2
  HGB: Unknown | 0 | 0 | 0 | 1
  HGB: Below | 22 | 22 | 27 | 23
  HGB: Normal | 8 | 7 | 4 | 6
  HGB: Above | 0 | 0 | 0 | 0
  HCT: Unknown | 0 | 1 | 0 | 1
  HCT: Below | 23 | 21 | 27 | 25
  HCT: Normal | 7 | 7 | 4 | 4
  HCT: Above | 0 | 0 | 0 | 0
  LDH: Unknown | 0 | 0 | 1 | 0
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 28 | 28 | 29 | 27
  LDH: Above | 2 | 1 | 1 | 3
  LYM: Unknown | 0 | 0 | 0 | 1
  LYM: Below | 11 | 14 | 6 | 9
  LYM: Normal | 19 | 15 | 23 | 19
  LYM: Above | 0 | 0 | 2 | 1
  MON: Unknown | 0 | 0 | 0 | 1
  MON: Below | 3 | 4 | 1 | 2
  MON: Normal | 27 | 25 | 30 | 27
  MON: Above | 0 | 0 | 0 | 0
  NEU: Unknown | 0 | 0 | 0 | 1
  NEU: Below | 4 | 3 | 7 | 3
  NEU: Normal | 26 | 25 | 23 | 26
  NEU: Above | 0 | 1 | 1 | 0
  PLAT: Unknown | 0 | 0 | 0 | 1
  PLAT: Below | 2 | 6 | 6 | 10
  PLAT: Normal | 28 | 23 | 25 | 19
  PLAT: Above | 0 | 0 | 0 | 0
  PT: Unknown | 2 | 0 | 1 | 4
  PT: Below | 0 | 0 | 0 | 0
  PT: Normal | 27 | 28 | 30 | 25
  PT: Above | 1 | 1 | 0 | 1
  PTT: Unknown | 2 | 0 | 1 | 4
  PTT: Below | 0 | 1 | 0 | 0
  PTT: Normal | 27 | 24 | 27 | 22
  PTT: Above | 1 | 4 | 3 | 4
  RBC: Unknown | 0 | 1 | 0 | 1
  RBC: Below | 24 | 25 | 29 | 26
  RBC: Normal | 6 | 3 | 2 | 3
  RBC: Above | 0 | 0 | 0 | 0
  TP: Unknown | 0 | 0 | 0 | 0
  TP: Below | 5 | 3 | 8 | 7
  TP: Normal | 25 | 26 | 23 | 23
  TP: Above | 0 | 0 | 0 | 0
  WBC: Unknown | 0 | 0 | 0 | 1
  WBC: Below | 9 | 8 | 9 | 6
  WBC: Normal | 21 | 20 | 20 | 22
  WBC: Above | 0 | 1 | 2 | 1

9. Primary Outcome: Number of Subjects With Hematological and Biochemical Parameters With Respect to Normal Laboratory Ranges
Description: as for outcome 8
Time Frame: At Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 30 | 30
Participants
  ALT: Unknown | 0 | 0 | 1 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 26 | 28 | 29 | 27
  ALT: Above | 4 | 1 | 0 | 3
  AST: Unknown | 0 | 0 | 1 | 1
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 25 | 29 | 29 | 27
  AST: Above | 5 | 0 | 0 | 2
  BAS: Unknown | 0 | 1 | 1 | 0
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 30 | 28 | 29 | 30
  BAS: Above | 0 | 0 | 0 | 0
  CAL: Unknown | 0 | 0 | 1 | 1
  CAL: Below | 1 | 2 | 0 | 1
  CAL: Normal | 29 | 26 | 29 | 28
  CAL: Above | 0 | 1 | 0 | 0
  CREA: Unknown | 0 | 0 | 1 | 0
  CREA: Below | 0 | 0 | 0 | 0
  CREA: Normal | 29 | 27 | 26 | 27
  CREA: Above | 1 | 2 | 3 | 3
  EOS: Unknown | 0 | 1 | 1 | 0
  EOS: Below | 7 | 6 | 8 | 7
  EOS: Normal | 23 | 22 | 19 | 22
  EOS: Above | 0 | 0 | 2 | 1
  FIBR: Unknown | 0 | 1 | 0 | 1
  FIBR: Below | 3 | 2 | 0 | 5
  FIBR: Normal | 24 | 20 | 26 | 22
  FIBR: Above | 3 | 6 | 4 | 2
  HGB: Unknown | 0 | 1 | 1 | 0
  HGB: Below | 19 | 18 | 23 | 25
  HGB: Normal | 11 | 10 | 6 | 5
  HGB: Above | 0 | 0 | 0 | 0
  HCT: Unknown | 0 | 1 | 1 | 0
  HCT: Below | 22 | 19 | 24 | 25
  HCT: Normal | 8 | 9 | 5 | 5
  HCT: Above | 0 | 0 | 0 | 0
  LDH: Unknown | 0 | 0 | 1 | 1
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 30 | 28 | 29 | 27
  LDH: Above | 0 | 1 | 0 | 2
  LYM: Unknown | 0 | 1 | 1 | 0
  LYM: Below | 11 | 13 | 8 | 9
  LYM: Normal | 19 | 15 | 21 | 21
  LYM: Above | 0 | 0 | 0 | 0
  MON: Unknown | 0 | 1 | 1 | 0
  MON: Below | 8 | 5 | 2 | 5
  MON: Normal | 22 | 22 | 27 | 25
  MON: Above | 0 | 1 | 0 | 0
  NEU: Unknown | 0 | 1 | 1 | 0
  NEU: Below | 6 | 9 | 5 | 6
  NEU: Normal | 24 | 19 | 24 | 23
  NEU: Above | 0 | 0 | 0 | 1
  PLAT: Unknown | 0 | 1 | 1 | 1
  PLAT: Below | 5 | 4 | 5 | 7
  PLAT: Normal | 25 | 24 | 24 | 22
  PLAT: Above | 0 | 0 | 0 | 0
  PT: Unknown | 0 | 1 | 0 | 1
  PT: Below | 0 | 0 | 0 | 0
  PT: Normal | 28 | 25 | 29 | 28
  PT: Above | 2 | 3 | 1 | 1
  PTT: Unknown | 0 | 1 | 0 | 1
  PTT: Below | 0 | 1 | 0 | 0
  PTT: Normal | 26 | 23 | 26 | 26
  PTT: Above | 4 | 4 | 4 | 3
  RBC: Unknown | 0 | 1 | 1 | 0
  RBC: Below | 24 | 24 | 25 | 29
  RBC: Normal | 6 | 4 | 4 | 1
  RBC: Above | 0 | 0 | 0 | 0
  TP: Unknown | 0 | 0 | 1 | 0
  TP: Below | 3 | 2 | 6 | 6
  TP: Normal | 27 | 27 | 23 | 24
  TP: Above | 0 | 0 | 0 | 0
  WBC: Unknown | 0 | 1 | 1 | 0
  WBC: Below | 13 | 10 | 8 | 13
  WBC: Normal | 17 | 17 | 21 | 16
  WBC: Above | 0 | 1 | 0 | 1

10. Primary Outcome: Number of Subjects With Hematological and Biochemical Parameters With Respect to Normal Laboratory Ranges
Description: as for outcome 8
Time Frame: At Month 2
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 28 | 29 | 28
Participants
  ALT: Unknown | 1 | 1 | 0 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 26 | 26 | 29 | 24
  ALT: Above | 3 | 1 | 0 | 4
  AST: Unknown | 1 | 1 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 28 | 26 | 29 | 26
  AST: Above | 1 | 1 | 0 | 2
  BAS: Unknown | 1 | 0 | 0 | 1
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 29 | 28 | 29 | 27
  BAS: Above | 0 | 0 | 0 | 0
  CAL: Unknown | 1 | 1 | 0 | 0
  CAL: Below | 1 | 0 | 0 | 0
  CAL: Normal | 27 | 26 | 28 | 27
  CAL: Above | 1 | 1 | 1 | 1
  CREA: Unknown | 1 | 1 | 0 | 0
  CREA: Below | 0 | 0 | 0 | 0
  CREA: Normal | 28 | 25 | 26 | 25
  CREA: Above | 1 | 2 | 3 | 3
  EOS: Unknown | 1 | 0 | 0 | 1
  EOS: Below | 7 | 7 | 5 | 1
  EOS: Normal | 21 | 21 | 22 | 25
  EOS: Above | 1 | 0 | 2 | 1
  FIBR: Unknown | 1 | 1 | 0 | 1
  FIBR: Below | 4 | 0 | 4 | 4
  FIBR: Normal | 23 | 24 | 23 | 21
  FIBR: Above | 2 | 3 | 2 | 2
  HGB: Unknown | 1 | 0 | 0 | 1
  HGB: Below | 17 | 15 | 20 | 19
  HGB: Normal | 12 | 13 | 9 | 8
  HGB: Above | 0 | 0 | 0 | 0
  HCT: Unknown | 1 | 0 | 0 | 1
  HCT: Below | 20 | 18 | 21 | 21
  HCT: Normal | 9 | 10 | 8 | 6
  HCT: Above | 0 | 0 | 0 | 0
  LDH: Unknown | 1 | 1 | 0 | 0
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 28 | 24 | 29 | 26
  LDH: Above | 1 | 3 | 0 | 2
  LYM: Unknown | 1 | 0 | 0 | 1
  LYM: Below | 10 | 14 | 4 | 5
  LYM: Normal | 19 | 14 | 25 | 22
  LYM: Above | 0 | 0 | 0 | 0
  MON: Unknown | 1 | 0 | 0 | 1
  MON: Below | 4 | 5 | 2 | 5
  MON: Normal | 24 | 23 | 27 | 22
  MON: Above | 1 | 0 | 0 | 0
  NEU: Unknown | 1 | 0 | 0 | 1
  NEU: Below | 6 | 4 | 6 | 3
  NEU: Normal | 23 | 23 | 23 | 24
  NEU: Above | 0 | 1 | 0 | 0
  PLAT: Unknown | 1 | 0 | 0 | 1
  PLAT: Below | 3 | 4 | 5 | 7
  PLAT: Normal | 26 | 24 | 24 | 20
  PLAT: Above | 0 | 0 | 0 | 0
  PT: Unknown | 1 | 1 | 0 | 1
  PT: Below | 0 | 0 | 1 | 0
  PT: Normal | 27 | 25 | 28 | 26
  PT: Above | 2 | 2 | 0 | 1
  PTT: Unknown | 1 | 1 | 0 | 1
  PTT: Below | 0 | 0 | 1 | 0
  PTT: Normal | 23 | 22 | 24 | 25
  PTT: Above | 6 | 5 | 4 | 2
  RBC: Unknown | 1 | 0 | 0 | 1
  RBC: Below | 22 | 19 | 24 | 22
  RBC: Normal | 7 | 9 | 5 | 5
  RBC: Above | 0 | 0 | 0 | 0
  TP: Unknown | 1 | 1 | 0 | 0
  TP: Below | 2 | 1 | 4 | 3
  TP: Normal | 27 | 26 | 25 | 25
  TP: Above | 0 | 0 | 0 | 0
  WBC: Unknown | 1 | 0 | 0 | 1
  WBC: Below | 9 | 9 | 7 | 6
  WBC: Normal | 20 | 18 | 22 | 21
  WBC: Above | 0 | 1 | 0 | 0

11. Primary Outcome: Number of Subjects With Hematological and Biochemical Parameters With Respect to Normal Laboratory Ranges
Description: as for outcome 8
Time Frame: At Month 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 28 | 27 | 28 | 29
Participants
  ALT: Unknown | 0 | 0 | 1 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 25 | 26 | 27 | 27
  ALT: Above | 3 | 1 | 0 | 2
  AST: Unknown | 0 | 0 | 1 | 0
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 27 | 26 | 27 | 28
  AST: Above | 1 | 1 | 0 | 1
  BAS: Unknown | 3 | 1 | 0 | 1
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 25 | 26 | 28 | 27
  BAS: Above | 0 | 0 | 0 | 1
  CAL: Unknown | 0 | 0 | 1 | 0
  CAL: Below | 1 | 0 | 0 | 2
  CAL: Normal | 27 | 27 | 26 | 26
  CAL: Above | 0 | 0 | 1 | 1
  CREA: Unknown | 0 | 0 | 1 | 0
  CREA: Below | 0 | 0 | 0 | 0
  CREA: Normal | 28 | 25 | 24 | 26
  CREA: Above | 0 | 2 | 3 | 3
  EOS: Unknown | 3 | 1 | 0 | 1
  EOS: Below | 4 | 5 | 4 | 5
  EOS: Normal | 20 | 21 | 22 | 20
  EOS: Above | 1 | 0 | 2 | 3
  FIBR: Unknown | 1 | 0 | 0 | 0
  FIBR: Below | 1 | 3 | 3 | 4
  FIBR: Normal | 20 | 21 | 21 | 24
  FIBR: Above | 6 | 3 | 4 | 1
  HGB: Unknown | 3 | 1 | 0 | 1
  HGB: Below | 11 | 13 | 14 | 18
  HGB: Normal | 14 | 13 | 14 | 10
  HGB: Above | 0 | 0 | 0 | 0
  HCT: Unknown | 3 | 1 | 0 | 1
  HCT: Below | 13 | 15 | 20 | 18
  HCT: Normal | 12 | 11 | 8 | 10
  HCT: Above | 0 | 0 | 0 | 0
  LDH: Unknown | 0 | 0 | 1 | 0
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 28 | 27 | 27 | 27
  LDH: Above | 0 | 0 | 0 | 2
  LYM: Unknown | 3 | 1 | 0 | 1
  LYM: Below | 9 | 13 | 7 | 10
  LYM: Normal | 16 | 13 | 21 | 18
  LYM: Above | 0 | 0 | 0 | 0
  MON: Unknown | 3 | 1 | 0 | 1
  MON: Below | 2 | 6 | 2 | 5
  MON: Normal | 23 | 20 | 26 | 23
  MON: Above | 0 | 0 | 0 | 0
  NEU: Unknown | 3 | 1 | 0 | 1
  NEU: Below | 3 | 3 | 6 | 5
  NEU: Normal | 21 | 21 | 22 | 23
  NEU: Above | 1 | 2 | 0 | 0
  PLAT: Unknown | 3 | 2 | 0 | 1
  PLAT: Below | 2 | 3 | 5 | 8
  PLAT: Normal | 23 | 22 | 23 | 20
  PLAT: Above | 0 | 0 | 0 | 0
  PT: Unknown | 1 | 0 | 0 | 0
  PT: Below | 0 | 0 | 1 | 0
  PT: Normal | 25 | 25 | 27 | 27
  PT: Above | 2 | 2 | 0 | 2
  PTT: Unknown | 1 | 0 | 0 | 0
  PTT: Below | 0 | 0 | 1 | 0
  PTT: Normal | 20 | 23 | 22 | 25
  PTT: Above | 7 | 4 | 5 | 4
  RBC: Unknown | 3 | 1 | 0 | 1
  RBC: Below | 15 | 17 | 22 | 24
  RBC: Normal | 10 | 9 | 6 | 4
  RBC: Above | 0 | 0 | 0 | 0
  TP: Unknown | 0 | 0 | 1 | 0
  TP: Below | 2 | 3 | 3 | 4
  TP: Normal | 26 | 24 | 24 | 24
  TP: Above | 0 | 0 | 0 | 1
  WBC: Unknown | 3 | 1 | 0 | 1
  WBC: Below | 8 | 9 | 7 | 7
  WBC: Normal | 16 | 17 | 21 | 21
  WBC: Above | 1 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects With Hematological and Biochemical Parameters With Respect to Normal Laboratory Ranges
Description: as for outcome 8
Time Frame: At Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 29 | 26 | 27 | 26
Participants
  ALT: Unknown | 1 | 0 | 0 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 26 | 26 | 27 | 25
  ALT: Above | 2 | 0 | 0 | 1
  AST: Unknown | 1 | 1 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 28 | 25 | 27 | 24
  AST: Above | 0 | 0 | 0 | 2
  BAS: Unknown | 1 | 0 | 0 | 0
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 28 | 26 | 27 | 26
  BAS: Above | 0 | 0 | 0 | 0
  CAL: Unknown | 1 | 0 | 0 | 0
  CAL: Below | 3 | 0 | 0 | 1
  CAL: Normal | 25 | 26 | 27 | 25
  CAL: Above | 0 | 0 | 0 | 0
  CREA: Unknown | 1 | 0 | 0 | 0
  CREA: Below | 0 | 0 | 0 | 0
  CREA: Normal | 27 | 23 | 25 | 25
  CREA: Above | 1 | 3 | 2 | 1
  EOS: Unknown | 1 | 0 | 0 | 0
  EOS: Below | 3 | 4 | 3 | 2
  EOS: Normal | 24 | 21 | 23 | 22
  EOS: Above | 1 | 1 | 1 | 2
  FIBR: Unknown | 0 | 1 | 0 | 0
  FIBR: Below | 4 | 3 | 2 | 4
  FIBR: Normal | 16 | 19 | 22 | 22
  FIBR: Above | 9 | 3 | 3 | 0
  HGB: Unknown | 0 | 0 | 0 | 0
  HGB: Below | 17 | 11 | 14 | 20
  HGB: Normal | 12 | 15 | 13 | 6
  HGB: Above | 0 | 0 | 0 | 0
  HCT: Unknown | 0 | 0 | 0 | 0
  HCT: Below | 18 | 14 | 17 | 20
  HCT: Normal | 11 | 12 | 10 | 6
  HCT: Above | 0 | 0 | 0 | 0
  LDH: Unknown | 1 | 1 | 0 | 0
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 26 | 24 | 26 | 25
  LDH: Above | 2 | 1 | 1 | 1
  LYM: Unknown | 1 | 0 | 0 | 0
  LYM: Below | 7 | 10 | 9 | 6
  LYM: Normal | 21 | 16 | 18 | 19
  LYM: Above | 0 | 0 | 0 | 1
  MON: Unknown | 1 | 0 | 0 | 0
  MON: Below | 6 | 2 | 4 | 5
  MON: Normal | 22 | 24 | 23 | 21
  MON: Above | 0 | 0 | 0 | 0
  NEU: Unknown | 1 | 0 | 0 | 0
  NEU: Below | 4 | 2 | 7 | 4
  NEU: Normal | 23 | 24 | 20 | 22
  NEU: Above | 1 | 0 | 0 | 0
  PLAT: Unknown | 0 | 0 | 0 | 0
  PLAT: Below | 4 | 5 | 6 | 9
  PLAT: Normal | 25 | 21 | 21 | 17
  PLAT: Above | 0 | 0 | 0 | 0
  PT: Unknown | 0 | 1 | 0 | 0
  PT: Below | 0 | 0 | 1 | 0
  PT: Normal | 27 | 23 | 26 | 23
  PT: Above | 2 | 2 | 0 | 3
  PTT: Unknown | 0 | 1 | 0 | 0
  PTT: Below | 0 | 0 | 1 | 0
  PTT: Normal | 27 | 22 | 20 | 20
  PTT: Above | 2 | 3 | 6 | 6
  RBC: Unknown | 0 | 0 | 0 | 0
  RBC: Below | 21 | 15 | 23 | 23
  RBC: Normal | 8 | 11 | 4 | 3
  RBC: Above | 0 | 0 | 0 | 0
  TP: Unknown | 1 | 0 | 0 | 0
  TP: Below | 3 | 1 | 1 | 3
  TP: Normal | 25 | 25 | 26 | 23
  TP: Above | 0 | 0 | 0 | 0
  WBC: Unknown | 1 | 0 | 0 | 0
  WBC: Below | 8 | 7 | 8 | 9
  WBC: Normal | 19 | 19 | 19 | 16
  WBC: Above | 1 | 0 | 0 | 1

13. Primary Outcome: Frequency of gE-specific Cluster of Differentiation 4 (CD4) T-cells Expressing at Least 2 Cytokines
Description: The analysis focused on CD4 T-cells expressing at least 2 cytokines among Interferon gamma [IFN-γ], Interleukin 2 [IL-2], Tumour Necrosis Factor alpha [TNF-α] and/or CD40 Ligand [CD40L] as determined by in vitro intracellular cytokine staining (ICS).
Time Frame: At Month 4
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented. Only subjects with results available were included in this analysis.
Measure: Mean (Standard Deviation); unit: gE-specific CD4+ T-cells/million T-cells
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 27 | 25 | 22 | 23
gE-specific CD4+ T-cells/million T-cells | 11963.56 (11655.09) | 8114.83 (9957.55) | 6974.97 (10437.53) | 96.15 (108.08)
Statistical Analysis 1: Comparison: GSK 1437173A F1 Group; The null hypothesis was H0: GSK 1437173A F1 Group/Placebo Group below (<) 1; Test type: Superiority — Criterion for superiority: The Lower Limit (LL) of the Confidence Interval (CI) of the ratio of geometric means, in terms of ceellular immune (CMI) response for GSK 1437173A F1 Group as compared to Placebo Group, is above (>) 2; p < 0.0001, Dunnett for multiple comparisons; Fold increase over Control = 32.31, 76.16% CI 2-sided [20.65 to 50.54]
Statistical Analysis 2: Comparison: Placebo-GSK 1437173A F1 Group; The null hypothesis was H0: Placebo-GSK 1437173A F1 Group/Placebo Group < 2; Test type: Superiority — Criterion for superiority: The Lower Limit (LL) of the Confidence Interval (CI) of the ratio of geometric means, in terms of CMI response for Placebo-GSK 1437173A F1 Group as compared to Placebo Group, is above (>) 2; p < 0.0001, Dunnett for multiple comparisons; Fold increase over Control = 9.51, 76.16% CI 2-sided [6.07 to 14.9]

14. Primary Outcome: Anti-glycoprotein E (Anti-gE) Geometric Mean Antibody Concentrations
Description: Concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and are presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Month 4
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 29 | 26 | 27 | 26
mIU/mL | 29192.9 [11004.7 to 77442.1] | 22503.0 [8432.7 to 60050.2] | 11064.6 [4361.2 to 28071.8] | 406.0 [244.2 to 674.9]
Statistical Analysis 1: Comparison: GSK 1437173A F1 Group; The null hypothesis was H0: GSK 1437173A 1 Group/Placebo Group < 1; Test type: Superiority — Criterion for superiority: The Lower Limit (LL) of the Confidence Interval (CI) of the ratio of geometric means, in terms of humoral response for GSK 1437173A F1 Group as compared to Placebo Group, is above (>) 3; p < 0.0001, Dunnett for multiple comparisons; Fold increase over Control = 74.41, 76.16% CI 2-sided [33.12 to 167.17]
Statistical Analysis 2: Comparison: Placebo-GSK 1437173A F1 Group; The null hypothesis was H0: Placebo-GSK 1437173A 1 Group/Placebo Group < 1; Test type: Superiority — Criterion for superiority: The Lower Limit (LL) of the Confidence Interval (CI) of the ratio of geometric means, in terms of humoral response for Placebo-GSK 1437173A F1 Group as compared to Placebo Group, is above (>) 3; p < 0.0001, Dunnett for multiple comparisons; Fold increase over Control = 42.20, 76.16% CI 2-sided [20.20 to 88.13]

15. Primary Outcome: Anti-gE Mean Antibody Concentrations
Description: Concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and are presented as mean concentrations, expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Month 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 29 | 26 | 27 | 26
mIU/mL | 131471.10 (169644.69) | 102106.14 (116349.94) | 63768.06 (100839.95) | 840.46 (1119.44)

16. Secondary Outcome: Frequency of CD4 T-cells Specific for Varicella Zoster Virus (VZV) Antigens
Description: as for outcome 13
Time Frame: At Months 0, 1, 2, 3, 4 and 15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: VZV specific CD4+ T-cells/million Tcells
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 28 | 27 | 28 | 24
VZV specific CD4+ T-cells/million Tcells
  At Month 0: number analyzed (Participants) | 26 | 22 | 28 | 24
  At Month 0 | 356.11 (519.79) | 449.31 (637.09) | 343.90 (381.20) | 273.91 (280.07)
  At Month 1: number analyzed (Participants) | 28 | 27 | 26 | 23
  At Month 1 | 636.10 (886.14) | 1205.59 (2680.05) | 303.70 (383.32) | 486.97 (652.18)
  At Month 2: number analyzed (Participants) | 27 | 22 | 27 | 24
  At Month 2 | 3818.03 (3773.74) | 4466.98 (7100.05) | 928.35 (1773.80) | 249.91 (243.82)
  At Month 3: number analyzed (Participants) | 25 | 22 | 24 | 22
  At Month 3 | 3488.70 (4130.59) | 3628.20 (6682.51) | 887.86 (1244.78) | 511.33 (909.03)
  At Month 4: number analyzed (Participants) | 24 | 24 | 21 | 22
  At Month 4 | 5359.40 (6486.90) | 4243.82 (6216.73) | 4481.70 (6761.94) | 279.35 (246.06)
  At Month 15: number analyzed (Participants) | 24 | 18 | 17 | 18
  At Month 15 | 3104.65 (3543.66) | 3298.68 (4326.74) | 2669.66 (3121.01) | 320.39 (337.72)

17. Secondary Outcome: Frequency of gE-specific Cluster of Differentiation 4 (CD4) T-cells Expressing at Least 2 Cytokines
Description: as for outcome 13
Time Frame: At Months 0, 1, 2, 3 and 15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: gE-specific CD4+ T-cells/million T-cells
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 28 | 27
gE-specific CD4+ T-cells/million T-cells
  At Month 0: number analyzed (Participants) | 27 | 27 | 28 | 27
  At Month 0 | 116.53 (180.53) | 145.97 (217.01) | 83.15 (90.39) | 97.48 (148.32)
  At Month 1: number analyzed (Participants) | 30 | 29 | 28 | 26
  At Month 1 | 856.69 (1551.94) | 1376.95 (3358.49) | 91.84 (118.22) | 133.85 (204.90)
  At Month 2: number analyzed (Participants) | 29 | 26 | 27 | 26
  At Month 2 | 8830.03 (9745.11) | 9128.95 (12539.86) | 1528.60 (3204.39) | 124.53 (160.24)
  At Month 3: number analyzed (Participants) | 28 | 24 | 25 | 25
  At Month 3 | 7111.22 (7755.09) | 8415.89 (12235.84) | 827.83 (1508.97) | 158.13 (180.84)
  At Month 15: number analyzed (Participants) | 26 | 18 | 18 | 18
  At Month 15 | 6865.36 (6557.75) | 5900.24 (7728.98) | 3859.68 (4771.08) | 71.03 (80.76)

18. Secondary Outcome: Varicella Zoster Virus (VZV)-Specific Geometric Mean Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Months 0, 1, 2, 3, 4 and 15
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 28 | 28 | 29 | 28
mIU/mL
  At Month 0: number analyzed (Participants) | 28 | 26 | 29 | 27
  At Month 0 | 570.1 [393.1 to 826.8] | 755.1 [479.2 to 1189.9] | 639.9 [397.5 to 1030.1] | 659.2 [496.9 to 874.4]
  At Month 1: number analyzed (Participants) | 26 | 26 | 28 | 28
  At Month 1 | 922.2 [575.6 to 1477.4] | 1017.3 [609.6 to 1697.7] | 562.4 [346.9 to 912.0] | 729.4 [512.0 to 1039.2]
  At Month 2: number analyzed (Participants) | 27 | 28 | 26 | 27
  At Month 2 | 4268.5 [2075.7 to 8777.9] | 4541.3 [2506.4 to 8228.2] | 702.4 [398.5 to 1238.0] | 523.5 [351.8 to 779.2]
  At Month 3: number analyzed (Participants) | 24 | 24 | 24 | 28
  At Month 3 | 3940.7 [1819.0 to 8537.5] | 4598.3 [2292.6 to 9222.8] | 558.2 [302.3 to 1030.6] | 632.7 [374.5 to 1068.8]
  At Month 4: number analyzed (Participants) | 27 | 24 | 24 | 24
  At Month 4 | 8484.1 [4190.6 to 17176.4] | 6223.4 [2893.7 to 13384.5] | 3196.6 [1532.2 to 6668.9] | 351.9 [207.9 to 595.7]
  At Month 15: number analyzed (Participants) | 23 | 21 | 21 | 21
  At Month 15 | 1946.5 [1013.4 to 3738.6] | 2598.2 [1327.4 to 5085.6] | 930.3 [390.1 to 2218.6] | 339.4 [159.0 to 724.1]

19. Secondary Outcome: VZV-specific Mean Antibody Concentrations
Description: Concentrations are presented as mean concentrations, expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Months 0, 1, 2, 3, 4 and 15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 28 | 28 | 29 | 28
mIU/mL
  At Month 0: number analyzed (Participants) | 28 | 26 | 29 | 27
  At Month 0 | 968.22 (1466.46) | 1340.29 (1685.09) | 1304.22 (1866.32) | 843.07 (616.78)
  At Month 1: number analyzed (Participants) | 26 | 26 | 28 | 28
  At Month 1 | 1881.91 (2742.85) | 1957.16 (2438.00) | 1089.57 (1586.68) | 1158.99 (1407.26)
  At Month 2: number analyzed (Participants) | 27 | 28 | 26 | 27
  At Month 2 | 15155.95 (22198.03) | 10934.78 (13735.35) | 1506.49 (2120.19) | 911.09 (1211.24)
  At Month 3: number analyzed (Participants) | 24 | 24 | 24 | 28
  At Month 3 | 13342.90 (19278.57) | 12602.99 (18030.89) | 1227.40 (1794.62) | 2902.89 (10461.29)
  At Month 4: number analyzed (Participants) | 27 | 24 | 24 | 24
  At Month 4 | 23858.74 (31173.45) | 16752.32 (17738.95) | 10744.24 (17397.97) | 753.59 (1155.17)
  At Month 15: number analyzed (Participants) | 23 | 21 | 21 | 21
  At Month 15 | 4694.74 (5945.23) | 5482.75 (5769.88) | 2956.21 (4515.53) | 835.21 (947.65)

20. Secondary Outcome: Anti-gE Geometric Mean Antibody Concentrations
Description: as for outcome 14
Time Frame: At Months 0, 1, 2, 3 and 15
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 28 | 30 | 30
mIU/mL
  At Month 0 | 531.2 [402.6 to 700.8] | 536.2 [304.0 to 945.7] | 448.0 [289.7 to 692.8] | 659.9 [470.5 to 925.4]
  At Month 1: number analyzed (Participants) | 30 | 28 | 30 | 29
  At Month 1 | 1489.7 [847.3 to 2619.0] | 1288.1 [684.9 to 2422.5] | 376.1 [239.7 to 590.1] | 619.3 [424.2 to 904.0]
  At Month 2: number analyzed (Participants) | 30 | 28 | 29 | 28
  At Month 2 | 11963.0 [4739.4 to 30196.6] | 11628.8 [5196.6 to 26022.8] | 1047.8 [564.8 to 1943.9] | 520.2 [349.3 to 774.8]
  At Month 3: number analyzed (Participants) | 28 | 27 | 28 | 29
  At Month 3 | 13412.9 [4967.1 to 36219.7] | 13385.4 [5506.5 to 32537.7] | 972.6 [520.6 to 1817.2] | 585.2 [310.0 to 1104.9]
  At Month 15: number analyzed (Participants) | 27 | 22 | 23 | 21
  At Month 15 | 8052.7 [3333.4 to 19453.7] | 9165.5 [3796.0 to 22130.1] | 2968.0 [1184.7 to 7436.1] | 362.3 [170.7 to 768.7]

21. Secondary Outcome: Anti-gE Mean Antibody Concentrations
Description: as for outcome 15
Time Frame: At Months 0, 1, 2, 3 and 15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 28 | 30 | 30
mIU/mL
  At Month 0 | 683.78 (501.88) | 1366.94 (2510.90) | 763.58 (818.71) | 1025.07 (1177.35)
  At Month 1: number analyzed (Participants) | 30 | 28 | 30 | 29
  At Month 1 | 4435.62 (7776.94) | 3812.19 (7197.49) | 675.39 (776.37) | 1016.00 (1159.33)
  At Month 2: number analyzed (Participants) | 30 | 28 | 29 | 28
  At Month 2 | 76302.68 (118526.31) | 47344.49 (78643.10) | 2951.78 (4785.22) | 927.04 (1221.66)
  At Month 3: number analyzed (Participants) | 28 | 27 | 28 | 29
  At Month 3 | 88592.39 (133279.24) | 62174.90 (94796.54) | 2739.11 (4458.45) | 8908.62 (42086.07)
  At Month 15: number analyzed (Participants) | 27 | 22 | 23 | 21
  At Month 15 | 42128.75 (66869.22) | 30938.91 (45130.79) | 16564.63 (30523.28) | 1091.74 (1585.07)

22. Secondary Outcome: Number of Subjects With Confirmed Herpes Zoster (HZ) Cases
Description: A suspected case of HZ could be confirmed by PCR and/or by clinical review of the GSK physician responsible for the study. Rash lesion samples collected from subjects clinically diagnosed as having a suspected case of HZ were tested by by polymerase chain reaction (PCR) using standardized and validated procedures for the laboratory diagnosis of HZ. If the PCR specimen was inadequate or was missing, suspected HZ cases were to be classified as 'a confirmed case of HZ' or 'not a case of HZ' based on the determination by the GSK responsible physician of the study.
Time Frame: During the entire study period (from Day 0 to Month 15)
Population: he analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
Number analyzed (Participants) | 30 | 29 | 31 | 30
Participants | 0 | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day post-vaccination period (Days 0-6); Unsolicited AEs: during the 30-day post-vaccination period (Days 0-29); SAEs: during the entire study period (Day 0 - Month 15).
Arm/Group | GSK 1437173A F1 Group | GSK 1437173A F2 Group | Placebo-GSK 1437173A F1 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 3/30 | 1/29 | 2/31 | 3/30
Serious Adverse Events (participants affected / at risk) | 6/30 | 9/29 | 10/31 | 8/30
Other Adverse Events (participants affected / at risk) | 29/30 | 27/29 | 29/31 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 1437173A F1 Group (N=30) | GSK 1437173A F2 Group (N=29) | Placebo-GSK 1437173A F1 Group (N=31) | Placebo Group (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Peripheral t-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 1437173A F1 Group (N=30) | GSK 1437173A F2 Group (N=29) | Placebo-GSK 1437173A F1 Group (N=31) | Placebo Group (N=30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 2 (2) | 1 (3) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 6 (10) | 7 (12) | 7 (10) | 1 (1)
Fatigue (General disorders) | 18 (39) | 18 (30) | 25 (44) | 10 (23)
Gastrointestinal disorder (Gastrointestinal disorders) | 10 (17) | 7 (11) | 11 (16) | 4 (6)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 13 (26) | 3 (3) | 12 (21) | 6 (8)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (46) | 18 (32) | 23 (41) | 8 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1) | 1 (1) | 3 (4)
Pain (General disorders) | 27 (73) | 22 (53) | 24 (49) | 7 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 12 (19) | 9 (11) | 12 (17) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Swelling (General disorders) | 6 (6) | 4 (5) | 4 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.